CLINICAL TRIAL: NCT02591641
Title: Use of a Shear Reduction Surface in Pre-hospital Transport
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ann N. Tescher,Ph.D., Clinical Nurse Specialist, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-004912
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Shear Strength
Keywords: pre-hospital transport; shear force; tissue interface pressure
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care First, then Liquicell (Experimental): Subjects were secured on a standard ambulance stretcher, with a shear and pressure sensors attached to the body. Starting at 0 degrees head-of-bed (HOB) elevation, the ambulance traveled on a closed driver training course accelerating up to 30 mph and decelerating to a stop 5 times. Shear and pressure measurements were taken during the runs. The HOB was then elevated to 15 and 30 degrees respectively, and the procedure repeated. Subjects were asked to rate their comfort at each of the HOB elevations using a 0-10 scale. Following the first set of 15 runs, the course was repeated with the LiquiCell® ASMO.
  Interventions: Device: Anti-shear mattress overlay; Other: Standard of Care
- Liquicell First, then Standard of Care (Experimental): Subjects were secured on a standard ambulance stretcher with an anti-shear mattress overlay placed on top of the stretcher, with a shear and pressure sensor attached to the body. Starting at 0 degrees head-of-bed (HOB) elevation, the ambulance traveled on a closed driver training course accelerating up to 30 mph and decelerating to a stop 5 times. Shear and pressure measurements were taken throughout the runs. The HOB was then elevated to 15 and 30 degrees respectively, and the procedure repeated. Subjects were asked to rate their comfort at each of the HOB elevations using a 0-10 scale. Following the first set of 15 runs, the course was repeated without the LiquiCell ASMO.
  Interventions: Device: Anti-shear mattress overlay; Other: Standard of Care

INTERVENTIONS:
Device: Anti-shear mattress overlay — A commercial full-length LiquiCell® anti-shear mattress overlay (ASMO) was placed on the standard ambulance stretcher mattress.
  Other Names: LiquiCell
Other: Standard of Care — Standard ambulance stretcher mattress

SUMMARY:
The purpose of this study was to examine the effectiveness of a shear reduction surface on shear, pressure, and comfort used in pre-hospital ground transport.

DETAILED DESCRIPTION:
This study enrolled healthy adult volunteers of any race or gender, stratified into 3 Body Mass Index (BMI) categories (≤20, 20.1-24.9, ≥25), who served as their own controls. The setting for this study was on a closed driving course utilized for training of emergency and law enforcement personnel, and the vehicle used was a standard ground ambulance affiliated with the Medical Transport of a tertiary medical center.

Apparatus and/or instruments: A commercial full-length LiquiCell® anti-shear mattress overlay (ASMO) (Birchwood Laboratories, Eden Prairie MN) was placed on the standard ambulance stretcher mattress. Shear force and tissue interface pressure was measured during a full stop, acceleration, travelling at 30 mph, deceleration, and a full stop by a PREDIA device (Molten Corporation, Hiroshima Japan) through reusable sensors attached to the sacrum, ischial tuberosity, and heel.

Procedures: Following written informed consent, subjects were weighed and measured with a calibrated scale to calculate a current BMI. Three PREDIA sensors were secured to three sites (sacrum, ischial tuberosity, and heel) with double-stick tape. Subjects wore standard hospital scrub bottoms, and were secured supine to the ambulance stretcher using standard procedure. Subjects were blinded to the presence of the LiquiCell® ASMO overlay by a sheet covering on the stretcher. The ASMO was placed according to a simple randomization table. The stretcher was initially be placed with 0 degree head-of-bed (HOB) elevation, followed by subsequent HOB elevations of 15 degrees and 30 degrees. HOB elevations were verified using a standard goniometer. The ambulance traveled over a closed course driven by ambulance staff members that had passed the mandatory Coaching the Emergency Vehicle Operator (CEVO) driving course. The course included at maximum speed of 30 mph and 5 complete stops at each of 3 HOB elevations (0, 15, and 30 degrees). Shear measurements (measured in Newtons) and pressure measurements (measured in mmHg) for each anatomical site were taken with the PREDIA sensors during a full stop, acceleration, travelling at 30 mph, deceleration, and a full stop for each "run". At the beginning and completion of each set of 5 runs, subjects were asked to rate their discomfort on a scale of 0 (no discomfort) to 10 (worst discomfort imaginable). Following the first set of 15 runs, the course was repeated with or without the LiquiCell® ASMO according to the randomization table.

ELIGIBILITY:
Inclusion criteria:

* Healthy adult volunteers
* 18-70 years old
* Able to read and write English
* Height of 6' feet tall or less
* Weight under 300 lbs.

Exclusion criteria:

* Non-English speaking
* Pregnancy
* Prisoners
* Previous history of pelvic fracture, pressure ulcers on sacrum, ischial tuberosity, or heel
* Adhesive allergy or sensitivity
* Height over 6 feet tall
* Weight over 300 lbs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Shear Force as as measured by the PREDIA monitor | baseline, 2 hours
  The PREDIA monitor is a hand-held monitor that measures both shear forced (measured in Newtons) and tissue-interface pressure (measured in mmHg) simultaneously at discrete points in time.

SECONDARY OUTCOMES:
Change in Tissue-Interface Pressure as measured by the PREDIA monitor | baseline, 2 hours
  The PREDIA monitor is a hand-held monitor that measures both shear forced (measured in Newtons) and tissue-interface pressure (measured in mmHg) simultaneously at discrete points in time.
Change in Comfort Score | baseline, 2 hours
  At the beginning and completion of each set of 5 runs, subjects were asked to rate their discomfort on a scale of 0 (no discomfort) to 10 (worst discomfort imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Ann Tescher, APRN, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No